CLINICAL TRIAL: NCT03797352
Title: HOPE (Healthy Older People Everyday) To Age in Place: Design and Implementation of an Innovative and Cost Effective Electronic Rapid Geriatric Assessment Tool for the Screening and Management of Frailty in Community Dwelling Older Adults
Brief Title: HOPE (Healthy Older People Everyday) To Age in Place
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Medicine, Head & Senior Consultant, Division of Geriatric Medicine, National University Hospital, Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2108/11
Record Dates: First submitted 2019-01-01; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Frail Elderly Syndrome
Keywords: Bone Health; Cognitive Decline; Health Education; Mobility Decline
MeSH Terms: conditions — Cognitive Dysfunction; Health Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receive healthy ageing advice every 3 months for the duration of 12 months
- Intervention (Experimental): To participate in supervised Multicomponent exercise (combined exercise and cognitive activity) up to three times a week for 6 months and receive healthy ageing advice
  Interventions: Other: Multicomponent exercise

INTERVENTIONS:
Other: Multicomponent exercise — To identify frailty and other potential health issues, and determine if Multicomponent exercise helps at-risk elderly to have better health outcomes.
  Arms: Intervention

SUMMARY:
Certain clinical syndromes eg frailty, sarcopenia, dementia, depression, cognitive impairment, vision impairment, falls in older adults carry an increased risk for poor health outcomes and if identified early, can be prevented, delayed or reversible. There is evidence to suggest that exercise and dietary intervention can help delay or prevent sarcopenia, frailty and dementia. Through early screening and detection of frailty and cognitive impairment, the investigators will be able to identify participants at risk of future physical or mental decline in primary care setting and ambulatory care clinics. Those prefrail, frail but ambulant with / without cognitive impairment will be randomised to dual task exercise with/without cognitive stimulation therapy and health education. The main hypothesis is that the combination of multicomponent group exercise activities and dual task exercise is effective in reversing frailty and improving cognition.

DETAILED DESCRIPTION:
Major challenges in the Singapore healthcare landscape include a rapidly aging population, due to rising life expectancy at birth combined with declining total fertility, and an epidemiological transition in the main source of disease burden from communicable and infectious conditions to non-communicable, chronic conditions. While acute care will always remain a crucial component of healthcare delivery systems, the increased healthcare burden centered on chronic diseases and the concomitant aging population is putting increased strain on healthcare resources. Frailty is reversible and progression to dementia can be delayed. From most recent study, prevalence of pre-frailty is 37% and mild cognitive impairment about 15-20%. WHO's definition of healthy ageing is maintaining functional ability. Cognicise, a dual task exercise has shown to delay decline in cognition and there are many studies which shows aerobic exercise improves endurance. Patients seen in Geriatric, Medicine Clinic or polyclinics who are prefrail, frail but ambulant with / without cognitive impairment will be randomised to dual task exercise with/without cognitive stimulation therapy and health education. In addition, high protein diet has been shown to improve muscle protein synthesis. Therefore, the aims of the study are to assess: a) Assess the effectiveness of dual task exercise with/without cognitive stimulation therapy b) Effect of health education alone for delaying the progression to dementia and mobility decline c) Assess impact of exercise on inflammatory and bone health biomarkers eg IL, TNF, Osteocalcin, sclerostin and C telopeptide in a subgroup of older adults randomly selected.

ELIGIBILITY:
Inclusion Criteria:

* Pre frail or frail but ambulant (Frail scale score of at least 1)
* Able to walk 400m aided or unaided (at least one bus stop away)
* Has no significant heart or lung problems
* Grip strength not more than 25kg for males and 18kg for females

Exclusion Criteria:

* Unable to give consent personally
* Wheelchair bound or at a very high falls risk
* Unable to participate due to underlying health problems including severe weakness due to stroke
* Undergoing active cancer treatment

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Changes in frailty status | 1 year
  Changes in frailty status by 5-item FRAIL scale Scale range from 0 to 5, the higher the value, the more frail (3 or greater = frailty; 1 or 2 = prefrail)
Functional improvement | 1 year
  Changes in short physical performance battery (SPPB) summary score 3 subscales (range from 0 to 4 for balance, gait speed and chair stand) summed to give total score range from 0 to 12. The higher the value, the better the performance of lower extremity.

SECONDARY OUTCOMES:
Upper extremity strength | 1 year
  Changes in handgrip strength test performance (kg)
Reduction of prevalence of depression | 1 year
  Changes in Geriatric Depression Scale (GDS) Scale range from 0 to 15, the higher the score, the greater the likelihood of depression. A score > 5 points is suggestive of depression, a score ≥ 10 points is almost always indicative of depression
reduction in social isolation | 1 year
  Changes in Lubben Social Network Scale (LSNS-6). Scale range from 0 to 30, the lower the value, the more likelihood of social isolation, A score of 12 and lower delineates "at-risk" for social isolation
Improved quality of life | 1 year
  Changes in EuroQoL-5D (EQ5D) score 5 subscales (1 to 5): Mobility, self-care, usual activities, pain/discomfort, anxiety/depressed Each subscale assessed individually.
Improved cognition | 1 year
  Changes in Montreal Cognitive Assessment (MoCA), the scoring range from 0 to 30, the lower the scoring, the more likelihood of cognitive impairment. A score of 26 and higher is generally considered normal.
Improved cognition | 1 year
  Changes in Mini Mental State Examination (MMSE) score 5 subscales: Orientation (0 to 10), Registration (0 to 3), Attention and Calculation (0 to 5), Recall (0 to 3), Language and Praxis (0 to 9). Total scale range from 0 to 30, the higher the value, the less cognitive impairment. A score of 23 or lower is indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Reshma Merchant, MD, Principal Investigator — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided